CLINICAL TRIAL: NCT01938287
Title: A Prospective, Open Label Study to Assess the 24-hour Intraocular Pressure Pattern Recorded With SENSIMED Triggerfish® in Healthy Subjects With Closed Eye
Brief Title: SENSIMED Triggerfish in Closed Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1301
Record Dates: First submitted 2013-07-26; First posted 2013-09-10 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish (Experimental)
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish

SUMMARY:
This study investigates the effect of eye opening/closure on the quality of IOP (intraocular pressure) related patterns recorded with SENSIMED Triggerfish. Each subject receives 2 24-hour recording sessions, one with the recorded eye open and the other with the eye closed,using an ophthalmic patch.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject without previous ophthalmic medical history (except from indication for glasses)
* Aged ≥18 years, of either sex
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The difference between start and end TF (SENSIMED Triggerfish) in a closed eye as compared to the difference between start to end TF in an open eye | 24 hours
  TF will be installed on subjects' eyes for 24 hours in two sessions. In one session the eye will remain open (except during sleep) while in the other session the eye will be closed using an ophthalmic patch throughout the 24 hours. For both sessions, the initial TF output value in millivolt equivalent will be subtracted from the final output value to yield the difference from start to end. The difference obtained in the session with closed eye will be divided by that of the session with open eye (ratio).

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Department of Ophthalmology, Glaucoma Sector, Geneva, Switzerland